CLINICAL TRIAL: NCT02741765
Title: Exercise and Transcranial Magnetic Stimulation: Increasing Brain Plasticity in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 15-00712
Record Dates: First submitted 2016-03-31; First posted 2016-04-18 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Parkinson Disease
Keywords: Transcranial Magnetic Stimulation; Exercise; Brain Plasticity
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Sham Group (Active Comparator): Sham group will receive Sham rTMS+Aerobic Exercise
  Interventions: Behavioral: Sham rTMS; Behavioral: Supervised aerobic exercise
- Group 2: Real Group (Experimental): rTMS+Aerobic Exercise
  Interventions: Other: Real rTMS; Behavioral: Supervised aerobic exercise

INTERVENTIONS:
Behavioral: Sham rTMS — Subjects will participate in daily sessions of sham-rTMS
  Arms: Group 1: Sham Group
Other: Real rTMS — Subjects will participate in a combination of rTMS
  Arms: Group 2: Real Group
Behavioral: Supervised aerobic exercise

SUMMARY:
This is a feasibility and exploratory study consisting of two parts: first, a cross-sectional (one-time) biomarker measurement comparing BDNF-TrkB (Brain-derived neurotrophic factor (BDNF) and its receptor, TrkB,) signaling and cortical plasticity in patients diagnosed with Parkinson's Disease (PD) vs. healthy controls matched by age. Second, a prospective, randomized, double blind trial of Transcranial Magnetic Stimulation (TMS) MAGSTIM Rapid2 Therapy System (TMS) (real or Sham) and aerobic exercise. This exploratory feasibility study will look at BDNF-TrkB signaling and cortical plasticity.

DETAILED DESCRIPTION:
Twenty-four PD patients (n=24) will be randomly assigned to receive one of two interventions for a duration of two weeks. In Group 1, subjects will participate in daily sessions of sham-rTMS followed by supervised aerobic exercise (Sham rTMS+Aerobic); in Group 2, subjects will participate in a combination of rTMS and supervised aerobic exercise (Real rTMS+Aerobic). Serum BDNF-TrkB signaling in lymphocytes and TMS-based electrophysiological measures of LTP-like plasticity will be measured. A comparison of such measures in a group of patients with PD and in a group of age-matched controls (n=12) will be analyzed to establish the effect of the disease on indices of plasticity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD according to the UK Brain Bank Criteria, confirmed by a neurologist with expertise in movement disorders;
* Hoehn and Yahr stage II to III;
* On a stable medication regimen since at least 2 weeks prior the enrolment in the study and, in the view of the treating neurologist, unlikely to require medication adjustments in the following 3-6 months.

Inclusion Criteria (Healthy Controls)

* Male or Female; aged 35-85

Exclusion Criteria (Healthy Controls)

* History of seizure disorder, including febrile seizures;
* Neurological disorder including PD, stroke, traumatic brain injury, fainting spells or syncope of unknown cause(s);
* Major or unstable medical illness;
* Pacemakers, neurostimulators, tattoos or metal foreign bodies in the head area (dental fillings are allowed);
* Untreated depression, or score of >20 on Beck Depression Inventory II;
* Taking any of the following medications within the six weeks prior to the start of the study: imipramine, amitriptyline, doxepin, nortriptyline, maprotiline, chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, theophylline, calcium channel blockers, beta blockers, tadalafil, vardenafil, avanafil, and sildenafil;
* Diagnosis of dementia, or Montreal Cognitive Assessment (MoCA) <20;
* Any clinically significant abnormality on vital signs
* Cardiopulmonary limitations: untreated high blood pressure, history of heart insufficiency (class II-III), coronary vascular disease, angina, arrhythmia, dyspnea on exertion and asthma

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-11; Primary Completion 2018-01-26 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
Recruitment Enrollment Numbers | 2 Weeks
Number of enrolled subjects that remain in study | 2 Weeks

SECONDARY OUTCOMES:
Plasticity measured by TMS-PAS25 (LTP-like plasticity biomarker) | 2 Weeks
  A paired associative paradigm at 25 ms (TMS-PAS-25) to quantify cortical LTP in M1 motor cortex will be used. As well as a repetitive biphasic magnetic stimulator (Magstim Rapid2 stimulator -Magstim Co., Whitland, U.K.) with a "Figure of eight" coil (outer diameters: 9 cm) and apply standard protocol for LTP-like measurements.
Measurements of lymphocytes | 2 Weeks
Measurements of TrkB | 2 Weeks
Measurements of serum BDNF | 2 Weeks
Timed Up and Go Test | 2 Weeks
Freezing of Gait Questionnaire (FOG-Q) | 2 Weeks
Parkinson's Disease Quality of Life (PDQ-39) | 2 Weeks
Parkinson's Disease Sleep Scale (PDSS) | 2 Weeks
Frontal Function Assessment (FAB) | 2 Weeks
LASA Physical Activity Questionnaire (LAPAQ) | 2 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Milton Biagioni, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States